CLINICAL TRIAL: NCT02728999
Title: Does Less Trendelenburg Make a Difference in Robotic Assisted Gynecological Procedures?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not want to expose additional subjects to Arterial Line placement
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHCIRB 5589 Trendelenburg
Record Dates: First submitted 2016-03-01; First posted 2016-04-06 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2018-01

CONDITIONS: Benign Female Reproductive System Neoplasm
Keywords: Trendelenburg position; Robotic assisted gynecologic procedures; benign gynecologic conditions
MeSH Terms: interventions — Vascular Access Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Steep Trendelenburg
  Interventions: Procedure: Steep Trendelenburg
- Group B (Experimental): Decreased Trendelenburg
  Interventions: Procedure: Decreased Trendelenburg

INTERVENTIONS:
Procedure: Steep Trendelenburg — •Subjects who undergo steep Trendelenburg will remain in 30 degrees of Trendelenburg, and the da Vinci robot will be docked.
  After subjects are asleep an arterial line will be place in one wrist by the anesthesiologist. It will be removed at the conclusion of the procedure.
  Other Names: Arterial Line in Wrist
  Arms: Group A
Procedure: Decreased Trendelenburg — •Subjects who undergo decreased Trendelenburg will be taken out of Trendelenburg to the minimal angle possible that enables adequate visualization, as determined by the primary surgeon, at which time robot will be docked.
  After subjects are asleep an arterial line will be place in one wrist by the anesthesiologist. It will be removed at the conclusion of the procedure.
  Other Names: Arterial Line in Wrist
  Arms: Group B

SUMMARY:
Patient/Population: Women over the age of 18, who are not pregnant and are undergoing benign, robotic-assisted gynecologic procedures at Lutheran General Hospital.

Intervention: Decreasing the angle of Trendelenburg for the procedure Control: Steep Trendelenburg, which is the usual standard of care, to the limit of the operative bed, which is 30 degrees.

Outcome: Outcomes will include the mean angle of Trendelenburg in the experimental arm and the difference in Trendelenburg between the two arms. Additional outcomes included will be end tidal Carbon dioxide, peak airway pressure, mean arterial pressure, heart rate and arterial Carbon dioxide. Secondary outcomes will include operative time, blood loss and conversion to laparotomy.

DETAILED DESCRIPTION:
For any patient undergoing robotic-assisted benign laparoscopic procedures at Lutheran General Hospital were eligible to participate. Each subject was randomized to steep or a decreased angle of Trendelenburg. While under anesthesia an arterial line would be placed to monitor vital signs. At specific time points throughout surgery, all vital signs were measured including End Tidal CO2, peak airway pressure, mean arterial pressure, heart rate and arterial CO2 as well as operative time, blood loss and conversion to laparotomy.

The arterial line was removed at the conclusion of the case, and all variables will be compared between the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* all women at Lutheran General Hospital undergoing robotic-assisted benign gynecologic procedures and who agree to participate in the study.
* Women who are 18 years or older on the day of surgery.
* Patients with any co-morbidity or prior surgery, as long as they are cleared by their surgeon and anesthesia to undergo robotic-assisted surgery.

Exclusion Criteria:

* pregnant women
* Anyone who is less than 18 years old on the day of surgery.
* Anyone who does not have the capacity to make independent medical decisions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
• Mean Angle of Trendelenburg during surgery (Degrees of the operative head down, measured by electronic angle meter) and the difference in the two arms | 0-240 minutes
  Measured using electronic Angle Meter from supine to Trendelenburg in degrees (0-30)

SECONDARY OUTCOMES:
Cardiovascular Outcomes- Heart rate | 0-240 minutes
  Heart rate (beats per minute) measured in beats per minute by anesthesiologist at the beginning of the case prior to insufflation, after insufflation, every 30 minutes while in Trendelenburg and at the end of the case.
Respiratory Parameter- arterial CO2 | 0-240 minutes
  Arterial CO2- Measured by taking an arterial blood gas from the arterial line by the anesthesiologist at the beginning of the case prior to insufflation, and then every hour while in Trendelenburg.
Respiratory Outcomes- End Tidal CO2 | 0-240 minutes
  End Tidal CO2 measured in mmHg by anesthesiologist at the beginning of the case prior to insufflation, after insufflation, every 30 minutes while in Trendelenburg and then at the end of the case.
Respiratory Outcomes- Peak Airway Pressure | 0-240 minutes
  Peak Airway Pressure (mm Hg) measured in mmHg by anesthesiologist at the beginning of the case prior to insufflation, after insufflation, every 30 minutes while in Trendelenburg and then at the end of the case.
Cardiovascular Outcomes- Mean arterial Pressure | 0-240 minutes
  Mean arterial pressure (mm hg) measured in mmHg by anesthesiologist at the beginning of the case prior to insufflation, after insufflation, every 30 minutes while in Trendelenburg and then at the end of the case.
Operative Time | 1-240 minutes
  The operative time will be measured (minutes) from the time the robot was docked until it is undocked.
Estimated Blood Loss | 0-240 minutes
  The blood loss (mL) will be measured by subtracting the irrigation fluid used from the fluid suctioned out during the procedure.
Redocking of the robot | 0-240 minutes
  It will be recorded whether the robot required undocking, placement in greater Trendelenburg and redocking of the robot in order to complete the procedure.
Conversion of surgical approach | 0-240 minutes
  It will be recorded whether the surgical approach was transitioned to traditional laparoscopy or laparotomy versus a robotic-assisted procedure as scheduled.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Sasaki, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Manuscript and conference presentation
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available starting 2/2018 for 6 months
Access Criteria: Any person that requests analyzed data.